CLINICAL TRIAL: NCT07348315
Title: Effectiveness of Apheresis Platelet-Rich Plasma Injection for Androgenic Alopecia: A Single-Arm Trial
Brief Title: Effectiveness of Apheresis Platelet-Rich Plasma Injection for Androgenic Alopecia
Acronym: PRP-AGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: zhang li (Other)
Responsible Party: Sponsor-Investigator, zhang li, Principal Investigator, The General Hospital of Western Theater Command
Organization: The General Hospital of Western Theater Command (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023xjsxxm-28
Record Dates: First submitted 2025-12-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Androgenic Alopecia
Keywords: Androgenetic Alopecia; Platelet-Rich Plasma
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Masking Description: To ensure objective assessment, all photographs were anonymized by removing any time or sequence identifiers. Subsequently, these photographs were randomly assigned to 2 or 3 independent, blinded physicians for the assessment of hair loss severity. The physicians were blinded to the treatment stage (before- or after-treatment), patient identity, and PRP cellular composition throughout the grading process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Apheresis PRP Injection (Experimental): All enrolled participants will receive autologous apheresis platelet-rich plasma (PRP) injections into the scalp according to the defined protocol. This is the only arm in this single-arm trial.
  Interventions: Biological: Autologous Apheresis PRP Injection

INTERVENTIONS:
Biological: Autologous Apheresis PRP Injection — Autologous PRP was prepared using a closed-system blood cell separator with disposable blood cell collection consumables, following the manufacturer's standardized protocol.
  Using a 30-gauge sterile needle, PRP was administered via intradermal and subcutaneous injections at multiple points across the treatment area, with an injection volume of 0.05 mL per point at intervals of approximately 0.5 cm.
  Participants received 3 to 5 sessions of autologous apheresis PRP injections into the scalp at intervals of 3-5 weeks.

SUMMARY:
This study was retrospectively registered. The goal of this single-arm, single-center, prospective clinical trial is to evaluate the effectiveness and safety of autologous apheresis platelet-rich plasma (PRP) injection in the treatment of androgenetic alopecia (AGA). The main questions it aims to answer are:

* Is apheresis PRP effective in improving hair growth outcomes in male patients with AGA?
* Is treatment response associated with key variables, including patient age, number of treatment sessions, baseline severity, and PRP cellular composition?
* Does PRP injection lead to any serious adverse events in the treatment of AGA? Researchers will record the effectiveness and adverse events following autologous apheresis PRP treatment for AGA and perform statistical analyses to evaluate treatment outcomes and their correlates with the variables of interest.

Participants will:

* Receive 3 to 5 sessions of autologous apheresis PRP injections into the scalp at intervals of 3-5 weeks.
* Have standardized photographs of the scalp taken from four angles (frontal, vertex, and bilateral sides) prior to each PRP injection.
* Attend a follow-up clinic visit or complete a telephone assessment one month after the final PRP injection.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is a progressive condition with limited optimal therapeutic options. While platelet-rich plasma (PRP) therapy has been explored, the apheresis technique offers a distinct method of PRP preparation that yields higher platelet purity and more consistent cellular composition compared to conventional centrifugation methods. This study is specifically designed to evaluate the clinical effectiveness of this autologous apheresis PRP and identify key predictors. Given the exploratory nature of this investigation aimed at generating preliminary efficacy and safety data for a specific PRP preparation method, a single-arm design was chosen.

The apheresis procedure was performed using a closed-system blood cell separator according to the manufacturer's standardized protocol. All injections were uniformly administered following a strict procedural guideline.

The primary endpoint, change in the BASP classification, was assessed by independent, blinded physicians. The associations between treatment response and key variables, including age, number of sessions, baseline severity, and PRP cellular composition were explored through correlation and regression models.

ELIGIBILITY:
Inclusion Criteria:

* History of hair loss for more than 6 months
* Diagnosed with androgenetic alopecia (AGA) based on the Chinese guideline for diagnosis and treatment of AGA
* In good general health with a body weight ≥ 50 kg
* No history of hypertension, diabetes, platelet dysfunction, or any other contraindication to PRP apheresis
* No use of finasteride, minoxidil, or any other treatment for hair loss within the 6 months preceding enrollment
* No recent use of glucocorticoids (topical to treatment site for 1 month; systemic for 2 weeks) prior to PRP apheresis
* No recent use of nonsteroidal anti-inflammatory drugs (within 48 hours) prior to PRP apheresis
* Blood tests within 2 weeks before PRP apheresis meeting the following criteria:

  1. Hemoglobin concentration > 120 g/L
  2. Hematocrit 0.30 to 0.50
  3. Platelet count > 110 × 10^9/L
  4. No clinically significant abnormalities in inflammation, coagulation, or electrolyte panels

Exclusion Criteria:

* Concurrent use of finasteride, minoxidil, or other hair growth treatments during the PRP treatment phase of the study
* Failure to complete a minimum of 3 consecutive PRP treatment sessions as per the study protocol
* Failure to complete the required follow-up assessments for any reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Response Based on the Basic and Specific (BASP) classification | Baseline (pre-first injection) and End of treatment (pre-final injection, ranging from Week 9 to Week 25)
  The proportion of participants achieving a positive response, defined as an improvement of at least one grade in either the Basic or Specific component of the BASP system, as assessed by blinded, independent physicians on standardized photographs after PRP treatment compared to baseline. As the protocol allows for 3 to 5 injection sessions at intervals of 3 to 5 weeks, the 'End of Treatment' visit occurs on a variable calendar date, falling between Week 9 and Week 25 after the first injection. This design ensures that the assessment captures the cumulative effect of the complete, individualized treatment course for each participant.

SECONDARY OUTCOMES:
Patient-Reported Improvement Questionnaire | At 1 month after treatment completion
  Patient-reported outcomes will be assessed using a four-item questionnaire covering hair quality, hair thickness, hair loss reduction, and overall satisfaction. Responses are recorded on a 3-point scale: -1 (deteriorated/dissatisfied), 0 (unchanged/neutral), +1 (improved/satisfied). The outcome will be reported as the proportion of participants reporting an improvement (score of +1) for each individual item.
Incidence of treatment-related adverse events. | From first treatment to 1 month after last treatment, up to 6 months
  The frequency and severity of all treatment-related adverse events that occur during the treatment and follow-up period. The incidence will be calculated as the number and percentage of participants experiencing at least one treatment-related adverse event, as well as the number of individual adverse event occurrences.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) underlying the results of this single-center, investigator-initiated trial are not publicly available due to restrictions in the informed consent documents, which do not explicitly permit public data sharing. Aggregated data supporting the main findings are available within the published article or from the corresponding author upon reasonable request.

DOCUMENTS (2):
  • Study Protocol (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT07348315/Prot_000.pdf
  • Informed Consent Form (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT07348315/ICF_001.pdf